CLINICAL TRIAL: NCT04799028
Title: Evaluation of Toddler Milk Containing L.Reuteri, Galacto-oligosaccharides and Palm-Oil Free Fat Blend On Bone Metabolism Among Healthy Toddlers
Brief Title: Evaluation of Toddler Milk Containing L.Reuteri, Galacto-oligosaccharides and Palm-Oil Free Fat Blend
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Société des Produits Nestlé (SPN) (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: 20.10.INF
Record Dates: First submitted 2021-03-11; First posted 2021-03-16 (Actual); Last update posted 2023-03-24 (Actual); Status verified 2023-03

CONDITIONS: Toddlers Bone Metabolism

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The study is a double-blinded study. The identity of specific product will be masked to subjects, support staff, investigators and sponsor's personnel except the manufacture and quality unit at Nestle (production factory).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Traditional children's fortified cow's milk (Active Comparator)
  Interventions: Other: Traditional cow's milk
- New toddler milk with synbiotics and fat blend (Experimental)
  Interventions: Other: Experimental milk
- Toddlers consuming habitual diet (Other)
  Interventions: Other: Habitual diet

INTERVENTIONS:
Other: Traditional cow's milk — Fortified cow's milk
  Arms: Traditional children's fortified cow's milk
Other: Experimental milk — Milk with synbiotics and fat blend
  Arms: New toddler milk with synbiotics and fat blend
Other: Habitual diet — Habitual diet
  Arms: Toddlers consuming habitual diet

SUMMARY:
The purpose of this study is to evaluate the effects of experimental growing up milk (EXPL) as compared to traditional children's fortified milk (CTRL) fed for 6 months on bone mass index.

DETAILED DESCRIPTION:
A randomized, double-blind controlled clinical trial was chosen to study the effects of toddler milk containing L. reuteri and GOS (4g/L) and a low sn-1, -3 fat blend when compared to a control formula. There is an additional unblinded habitual intake reference group (REF) for "real-world" comparison (including 58% non-dairy drinkers according to observational data).

ELIGIBILITY:
All subjects must comply with all the following criteria:

1. Written informed consent has been obtained from the parent(s)/legally acceptable representative (LAR).
2. Singleton, full-term gestational birth (≥ 37 completed weeks of gestation), with a birth weight of ≥ 2.5 kg and ≤ 4.5 kg.
3. Child is between 24 months ±1 week to 36 months ±1 week.
4. Child is not currently consuming nor has consumed any formulas or taking any supplements with pre- or probiotics at enrolment or in the past month.
5. Child's parent(s)/guardian is of legal age of consent, must understand the informed consent and other study documents, and is willing and able to fulfill the requirements of the study protocol.

All subjects presenting one or more of the following criteria are excluded from participation in the study:

1. Chronic infectious, metabolic, genetic illness or other disease including any condition that impacts feeding or growth.
2. History of bone, malabsorption, metabolic, congenital or chromosomal abnormality known to affect feeding or growth.
3. Use of systemic antibiotics or anti-mycotic medication in the 4 weeks preceding enrollment.
4. Known or suspected cows' milk protein intolerance / allergy, or lactose intolerance, or severe food allergies that impact diet.
5. Current breast milk feeding in place of all other milk, and/or milk alternatives.
6. Clinical signs of severe micronutrient deficiencies.
7. Parents not willing / not able to comply with the requirements of study protocol.
8. Child's participation in another interventional clinical trial.

Ages: 2 Years to 3 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 273 (Actual)
Dates: Start 2021-06-19 (Actual); Primary Completion 2022-08-16 (Actual); Study Completion 2022-10-28 (Actual)

PRIMARY OUTCOMES:
Speed of sound (SOS) | Day 1, Day 90, Day 180
  Speed of sound (SOS) using a quantitative ultrasound methods measured by Pediatric Sunlight 9000 device

SECONDARY OUTCOMES:
GI tolerance and stooling patterns | Day 1
  Stool patterns including stool frequency will be recorded retrospectively via 24-hour GI Symptom and Behavior Recall
GI tolerance and stooling patterns | Day 1
  Stool patterns including stool consistency will be recorded retrospectively via 24-hour GI Symptom and Behavior Recall
GI tolerance and stooling patterns | Day 90, Day 180
  Stool patterns including stool frequency will be recorded using 3-day GI Symptom and Behavior diary
GI tolerance and stooling patterns | Day 90, Day 180
  Stool patterns including stool consistency will be recorded using 3-day GI Symptom and Behavior diary
GI tolerance and stooling patterns | Day 1, Day 90, Day 180
  Parent perceptions of GI symptoms using parent-reported questionnaire Toddler Gut Comfort Questionnaire (GCQ) using VAS from 1-Never to 6-Always with higher scores indicating increasing GI burden.
GI tolerance and stooling patterns | Day 1, Day 90, Day 180
  Parent perceptions of GI-related behaviors using parent-reported questionnaire Toddler Gut Comfort Questionnaire (GCQ) using VAS from 1-Never to 6-Always with higher scores indicating increasing GI burden.
Stool analyses | Day 1, Day 180
  Excretion of fecal calcium fatty acid soaps
Stool analyses | Day 1, Day 180
  Measurement of stool calcium content
Serum vitamin D | Day 1, Day 180
  Measured by serum 25[OH]D concentration requiring 1mL of whole blood sample.
Urine and Blood bone turnover markers | Day 1, Day 180 (EXPL and CTRL groups only)
  Bone accretion markers in urinary [C-terminal cross-linked telopeptides of type I collagen (CTX)
Urine and Blood bone turnover markers | Day 1, Day 180 (EXPL and CTRL groups only
  serum procollagen type I N-terminal propeptide (PINP)
Gut microbiota | Day 1, Day 180
  Gut microbiota analyzed for microbiome composition and diversity using next generation shotgun metagenomics sequencing, requiring 3g of stool sample.
Stool analyses | Day 1, Day 180
  Determination of fecal short chain fatty acids (SCFAs)
Stool analyses | Day 1, Day 180
  Fecal pH and metabolism.
Stool analyses | Day 1, Day 180
  Fecal markers of gut health
Physical strength | Day 1, Day 180
  Hand grip test (Jamar hand dynamometer) tailored for toddlers will be used as previously described Bohannon et al Pediatric Physical Therapy 2017.
Vitamin B | Day 1, Day 180
  serum vitamin B concentration requiring 2 mL of whole blood sample.
Dietary intake patterns | Day 1, Day 180
  Intake patterns are assessed using parent-reported questionnaire Child Eating Behavior Questionnaire including variety of food groups consumed as well as behaviors rated from Never to Always.
Child quality of life using validated ITQOL SF-47 questionnaire | Day 1, Day 180
  assessed using the parent-reported questionnaires
Outdoor Playtime | Day 1 and Day 180
  Assessed using parent-reported questionnaire on Outdoor Playtime recording number of hours child spent outside.
Child temperament | Day 1, Day 180
  Children's Behavior Questionnaire (very short form), consisting of 36 questions and 3 scales on child temperament domains Surgency, Negative Affect and Effort Control with each question ranging 1-extremely untrue to 7- extremely true of parent observing various behaviors.

OTHER OUTCOMES:
Anthropometry | Day 1, Day 180
  Measurement of weight
Anthropometry | Day 1, Day 180
  Measurement of height
Anthropometry | Day 1, Day 180
  Measurement of head circumference
Safety endpoints | Day 1, Day 180 and follow up of 14 days after last intake of study products
  Standard AEs reporting for safety assessment

CONTACTS AND LOCATIONS:
Locations (1):
- Asian Foundation for Tropical Medicine, Inc., City of Muntinlupa, Philippines

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Bonnet N, Capeding MR, Siegwald L, Garcia-Garcera M, Desgeorges T, Tytgat HLP, Krattinger LF, Lebumfacil J, Phee LC, Moll JM, Gudjonsson A, Rodriguez-Garcia P, Baruchet M, Feige JN, Jankovic I, Chen Y, Egli D, Horcajada MN. A young child formula with Limosilactobacillus reuteri and GOS modulates gut microbiome and enhances bone and muscle development: a randomized trial. Nat Commun. 2025 Dec 12;17(1):237. doi: 10.1038/s41467-025-66930-2. PMID 41387706